CLINICAL TRIAL: NCT07315061
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Study to Evaluate the Efficacy and Safety of D-2570 in Subjects With Active Psoriatic Arthritis
Brief Title: A Phase II Study to Evaluate the Efficacy and Safety of D-2570 in Subjects With Active Psoriatic Arthritis
Acronym: D2570-204
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2570-204
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: PsA (Psoriatic Arthritis)
Keywords: PsA (Psoriatic Arthritis)
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- D-2570 (experimental arm 1) (Experimental): Subjects will be randomized in a 1:1:1 ratio to D-2570 (experimental arm 1), D-2570 (experimental arm 2), or placebo (control arm). They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.
  Subjects assigned to the placebo group (control arm) completed a 12-week control treatment period,they will then be randomized in a 1:1 ratio to D-2570 (experimental arm 1), D-2570 (experimental arm 2).They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.
  Interventions: Drug: D-2570
- D-2570 (experimental arm 2) (Experimental): Subjects will be randomized in a 1:1:1 ratio to D-2570 (experimental arm 1), D-2570 (experimental arm 2), or placebo (control arm). They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks. Subjects assigned to the placebo group (control arm) completed a 12-week control treatment period,they will then be randomized in a 1:1 ratio to D-2570 (experimental arm 1), D-2570 (experimental arm 2).They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.
  Interventions: Drug: D-2570
- placebo (Placebo Comparator): Subjects will be randomized in a 1:1:1 ratio to D-2570 (experimental arm 1), D-2570 (experimental arm 2), or placebo (control arm). They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks. Subjects assigned to the placebo group (control arm) completed a 12-week control treatment period,they will then be randomized in a 1:1 ratio to D-2570 (experimental arm 1), D-2570 (experimental arm 2).They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.
  Interventions: Drug: D-2570; Drug: Placebo

INTERVENTIONS:
Drug: D-2570 — Subjects will then be randomized in a 1:1:1 ratio to D-2570 or placebo . They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.Subjects assigned to the placebo group (control arm) completed a 12-week control treatment period,they will then be randomized in a 1:1 ratio to D-2570 (experimental arm 1), D-2570 (experimental arm 2).They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.
Drug: Placebo — Subjects will then be randomized in a 1:1:1 ratio to D-2570 or placebo . They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.Subjects assigned to the placebo group (control arm) completed a 12-week control treatment period,they will then be randomized in a 1:1 ratio to D-2570 (experimental arm 1), D-2570 (experimental arm 2).They will enter the study treatment period and take the assigned investigational product once daily for 12 consecutive weeks.
  Arms: placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled clinical trial. The target population is patients with active psoriatic arthritis. A total of 222 subjects are planned to be included.

DETAILED DESCRIPTION:
The study is divided into three groups, each will include 74 subjects. The primary difference among the three groups lay in the dosage and whether they were placebo groups or not. In other aspects, such as population selection, randomization, blinding and outcome evaluation (safety and efficacy), are consistent among the three groups.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily take part in the study after being fully informed, sign a written informed consent form (ICF), and agree to follow procedures specified in the study protocol;
2. Males and females, 18 to 70 years of age, inclusive at the time of signing of ICF;
3. Have had an psoriatic arthritis of ≥ 3 months in duration prior to signing of ICF;
4. Have had active arthritis, characterized by at least ≥3 tender joints (68 joint tenderness counts) and ≥3 swollen joints (66 joint swelling counts).

Exclusion Criteria:

1. History of infection as defined in the protocol;
2. Any of the medical diseases or disorders listed in the protocol;
3. Significant, uncontrolled or unstable disease in any organ.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-08-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving ACR20 at Week 12 of treatment. | Week 12
  Definition of ACR20：The number of tender joints and swollen joints both decreased by at least 20% compared with the baseline.

SECONDARY OUTCOMES:
Proportion of subjects achieving minimal disease activity at Week 12 of treatment; | Week 12
Proportion of subjects achieving very low disease activity at Week 12 of treatment; | Week 12
Plasma concentrations of D-2570 | 0-week 24
safety（AEs） | 0-week 24
  An Adverse Event (AE) is definedas any new untoward medicaloccurrence or worsening of a preexistingmedical condition in a clinicalinvestigation participant administeredstudy treatment and that does notnecessarily have a causal relationshipwith this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: yi liu, phD, Principal Investigator — West China School of Medicine
Locations (1):
- West China School of Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No